CLINICAL TRIAL: NCT03496233
Title: "Study to Investigate the Efficacy of Elbasvir/Grazoprevir Fixed-Dose Combination for 8 Weeks in G1b Treatment-Naïve, HCV-Infected Patients With Non-severe Fibrosis, With or Without Glucose Abnormalities - EGG 18"
Brief Title: Elbasvir/Grazoprevir Fixed-Dose Combination for 8 Weeks in G1b Treatment-Naïve, HCV-Infected Patients
Acronym: EGG-18
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Principal Investigator, Antonio Craxi, Full Professor of Gastroenterology, Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017- 003710 -58
Record Dates: First submitted 2018-02-16; First posted 2018-04-12 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Chronic HCV Hepatitis
MeSH Terms: interventions — elbasvir; grazoprevir; Tablets; elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients included (Experimental): All patients included will be treated with Elbasvir/grazoprevir for 8 weeks
  Interventions: Drug: Elbasvir 50 MG / Grazoprevir 100 MG Oral Tablet [Zepatier]

INTERVENTIONS:
Drug: Elbasvir 50 MG / Grazoprevir 100 MG Oral Tablet [Zepatier] — Treatment with EBR/GZR Fixed-Dose Combination for 8 Weeks in G1b Treatment-Naïve, HCV-Infected Patients, with non- severe fibrosis, with or without IR and/or DM

SUMMARY:
Antiviral treatment of G1b Treatment-Naïve HCV-Infected Patients, with non- severe fibrosis, with or without insulin resistance (IR) and/or diabetes mellitus (DM) with EBR/GZR Fixed-Dose Combination for 8 Weeks.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Intervention Model: Single Group Assignment Masking: Open Label Primary Purpose: Treatment

Seventy-five (75) treatment-naïve subjects with chronic HCV GT1b infection (without cirrhosis) with or without glucose abnormalities such as insulin resistance and or diabetes will be consecutively enrolled.

The investigators decided to include also patients with glucose abnormalities at baseline screening since data on these patients are scanty, and inclusion of this subgroup of patients better reflects the clinical practice. The study will consecutively enroll patients, without fixing a specific rule (e.g. sample allocation ratio) for recruitment of patients with and without glucose abnormalities. This will allow to evaluate the proportion of patients with and without glucose abnormalities at baseline (a useful approach to understand the impact of patients with glucose abnormalities in real life) and to perform explorative analyses to compare patients with or without glucose abnormalities according to SVR.

There will be one treatment group with EBV/GZR (50/100 mg) once daily without regards to food for 8 weeks.

EBV/GZR is manufactured as a 50/100 mg tablet for oral administration. Subjects will take 1 tablet daily without regards to food.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Male or female, age ≥ 18 years
* Chronic HCV infection (≥ 6 months) documented by prior medical history or liver biopsy, only genotype 1b virus. (Positive for anti HCV antibody, HCV RNA, or an HCV genotype)
* Treatment-naïve with no prior exposure to any IFN, RBV, or approved or experimental HCV-specific DAA
* Non severe fibrosis (F≤ 2) according to Metavir score if a biopsy was performed or elasticity measured by Fibroscan® lower than 9.5 kPa or Fibrotest® lower than 0.59 or Fibrometer® lower than 0.63 if Fibroscan® cannot be performed.
* Patients who are HBV core antibody positive. These patients should be monitored for hepatitis flare or HBV reactivation during HCV treatment and post treatment follow-up. Appropriate patient management for HBV infection as clinically indicated should be initiated as recommended by the European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol (2017).
* Females of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 prior to enrollment
* Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use 2 effective method(s) of contraception from at least two weeks prior to Day 1 through 14 days after the last dose of study drugs.
* A female subject who is not of reproductive potential is eligible without requiring the use of contraception. A female subjects who is not of reproductive potentials is defined as one who has either 1) reached natural menopause (defined as 12 months with no menses without an alternative medical cause), 2) 6 weeks post surgical bilateral oophorectomy with or without hysterectomy, or 3) bilateral tubal ligation.
* A male subject who is not of reproductive potential is eligible without requiring the use of contraception. A male subject who is not of reproductive potential is defined as: one who has undergone a successful vasectomy. A successful vasectomy is defined as: (1) microscopic documentation of azoospermia, or (2) a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post vasectomy.
* Lactating females must agree to discontinue nursing before starting study drug
* Subject must be of generally good health, with the exception of chronic HCV infection, and glucose abnormalities as determined by the Investigator
* Subject must be able to comply with the dosing instructions for study drug administration

Exclusion Criteria:

* Is under the age of legal consent, is mentally or legally incapacitated, has a history of a clinically significant psychiatric disorder which, in the opinion of the investigator, would interfere with the study procedures.
* Current or prior history of any of the following:

  * Clinically significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol; subjects currently under evaluation for a potentially clinically significant illness (other than HCV) are also excluded
  * Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug
  * History of decompensation (e.g., clinical ascites, encephalopathy, and/or variceal hemorrhage)
  * Solid organ transplantation (including hematopoietic stem cell transplants) other than kidney, cornea and hair.
  * Significant cardiac disease
  * Unstable psychiatric condition including hospitalization, suicidal attempt, and/or a period of disability as a result of their psychiatric illness within 2 years prior to Screening
  * Malignancy within the 5 years prior to Screening, with the exception of specific cancers that have been cured by surgical resection (e.g., basal cell skin cancer, etc.). Subjects under evaluation for possible malignancy are not eligible
  * Significant drug allergy (e.g., hepatotoxicity)
* Subject has the following laboratory parameters at Screening:

  * ALT > 10 x the upper limit of normal (ULN)
  * AST > 10 x ULN
  * Direct bilirubin > 1.5 x ULN
  * Platelets < 75,000/μL
  * Creatinine clearance < 50 mL/min as calculated by the Cockcroft-Gault equation
  * Hemoglobin < 10 g/dL
  * Albumin < 3 g/dL
  * INR > 1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regime affecting INR
* Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, alfa-1 antitrypsin deficiency, cholangitis)
* Infection with human immunodeficiency virus (HIV)
* HBsAg positive patients
* Clinically-relevant alcohol or drug abuse within 12 months of Screening.
* Use of any prohibited concomitant medication listed in the specific SmPC section.
* Known hypersensitivity to the study drug, the metabolites, or formulation excipient
* Is currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another study.
* (female) is pregnant, lactating, expecting to conceive or donate eggs, or is of childbearing potential and unwilling to commit to two methods of birth control throughout treatment and after the completion of all treatment (see Inclusion Criteria); or male subject is planning to impregnate or provide sperm donation or has a female sexual partner of childbearing potential and is unwilling to commit to using a two methods of birth control throughout treatment and after the completion of all treatment (see Inclusion Criteria).
* had a life-threatening SAE during the screening period.
* is a member or a family member of the investigational study staff or sponsor staff directly involved with this study.
* has evidence or history of chronic hepatitis not caused by HCV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, and autoimmune hepatitis.
* For subjects diagnosed with diabetes mellitus, documented HbA1c >8.5% (to exclude uncontrolled diabetes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of elbasvir/grazoprevir fixed dose combination for 8 weeks in genotype 1b treatment naive HCV infected patients. | at 12 weeks
  Proportion of subject with sustained viral response (SVR) 12 weeks after cessation of treatment in G1b treatment naive HCV infected patients, with non severe fibrosis, with or without IR and/or DM treated with elbasvir/grazoprevir fixed dose combination for 8 weeks.

SECONDARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability). | 12 weeks after cessation of treatment
  Number (percentage) of participants with treatment related adverse events.
Insulin resistance | 12 weeks
  • Assessments of insulin resistance were measured using HOMA-IR at baseline and follow-up week (FW)12

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Undecided